CLINICAL TRIAL: NCT02605434
Title: Phase 3 Multicenter Randomized Double-Blind, Double-dummy, Active-Controlled Study Comparing Efficacy/Safety of Gastric-retentive, Controlled-release Accordion Pill Carbidopa/Levodopa to Immediate Release in Fluctuating Parkinson's Patients
Brief Title: A Study to Assess the Safety and Efficacy of the of the Gastric-retentive AP-CD/LD in Advanced Parkinson's Patients
Acronym: Accordance
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Intec Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IN 11 004
Record Dates: First submitted 2015-11-05; First posted 2015-11-16 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2018-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Fluctuating Parkinson's Disease; Advanced Parkinson's Disease; Carbidopa; Levodopa; Accordion; Accordance
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AP-CD/LD (Experimental): Accordion Pill™ Carbidopa/Levodopa Capsule 50/400mg , b.i.d or t.i.d or Accordion Pill™ Carbidopa/Levodopa Capsule 50/500mg , b.i.d or t.i.d and Placebo IR Carbidopa/ levodopa
  Interventions: Drug: Accordion Pill™ Carbidopa/Levodopa; Drug: Placebo -AP-CD/LD
- SINEMET® (Active Comparator): IR Carbidopa/ levodopa tablets 25/100 mg at least 4 times a day and placebo AP-CD/LD
  Interventions: Drug: Sinemet®; Drug: Placebo- Sinemet

INTERVENTIONS:
Drug: Accordion Pill™ Carbidopa/Levodopa — AP-CD/LD capsule containing 50 mg carbidopa with 400 mg or 500 mg levodopa administered orally twice or 3 times a day
  Other Names: AP-CD/LD
  Arms: AP-CD/LD
Drug: Sinemet® — Sinemet® tables containing carbidopa and levodopa 25/100 mg will be administered orally at least 4 times a day according to patients need
  Other Names: IR Carbidopa/Levodopa
  Arms: SINEMET®
Drug: Placebo -AP-CD/LD — Placebo for AP-CD/LD capsule
  Arms: AP-CD/LD
Drug: Placebo- Sinemet — Placebo for Sinemet tables
  Arms: SINEMET®

SUMMARY:
The purpose of this study is to determine whether the gastric retentive Accordion Pill™ Carbidopa/Levodopa (AP-CD/LD) is more effective than the commercially available immediate release Carbidopa/Levodopa in reducing motor fluctuations such as "off time" in advanced Parkinson's Disease patients.

DETAILED DESCRIPTION:
A multi-center, global, randomized, double-blind, double-dummy, active-controlled, parallel-group study in adult subjects with fluctuating PD. The study will have 2 open label Titration periods of 6 weeks each prior to the double blind Maintenance period. In the open label periods all patients will be stabilized on the active comparator Sinemet® and then on AP-CD/LD. The double blind Maintenance period will be 13 weeks long.

ELIGIBILITY:
Main Inclusion Criteria:

1. Subjects must be approved for suitability by an Enrollment Approval Committee
2. Able and willing to give written (signed and dated) informed consent and adhere to visit schedule and available to complete the study
3. Men or women 30 years of age and higher at initial screening assessment. (For the 100 subjects who enter the Gastroscopy sub study, the age limits are 30-80 years of age, inclusive, at initial screening assessment)
4. Diagnosed with Parkinson's disease, consistent with UK brain bank criteria
5. Has a good response to Levodopa and is taking at least 4 doses of a Levodopa containing medication (or 3 doses of Rytary) per day during waking hours (not including nighttime long acting levodopa) at a stable dose for at least 28 days prior to initial screening assessment
6. Other Anti-PD treatment (such as dopamine agonists, selective MAO-B inhibitors, anticholinergic agents or Amantadine) are permitted if stable for at least 28 days prior to study entry and provided they are not anticipated to be changed during the course of the study
7. Total LD immediate release daily dose of 400 mg to 1300 mg or equivalent prior to initial screening assessment. Specifically for Rytary, doses up to 1755 mg daily are acceptable.
8. Able to complete a Hauser Home Diary and can tell the difference between "On" and "Off" time

   1. Achieved at least 75% diary concordance with an approved site rater in a 4-hour training session including at least one "Off time" assessment
   2. Returned a valid 2-day practice diary after training has been completed.
9. At least 2.5 hours "Off time" per day during waking hours on Screening 2-day Practice Hauser Home Diary (morning akinesia should be incorporated into the total "Off time" assessment).
10. Other than PD, the subject is in satisfactory health, as assessed by physical examination and screening tests. No clinically significant medical, psychiatric or laboratory abnormality that could compromise safety or interfere with study procedures in the opinion of either the investigator or the Enrollment Approval Committee/Sponsor.
11. Living in an area that is within 3 hours driving distance from the study site or is willing to stay in such a place the night before each study visit

Main Exclusion Criteria:

1. Participation in another drug clinical trial within 28 days prior to initial screening assessment (calculated from the previous study's last dosing date)
2. Atypical Parkinsonism (subjects with Parkinsonian features caused by disorder such as multiple system atrophy, progressive supranuclear palsy, dementia with Lewy bodies or multiple brain infarcts)
3. Clinically significant cardiac, pulmonary, hepatic or renal disease or other condition or any major complication/illness which contraindicates his/her participation in the opinion of either the investigator or the Enrollment Approval Committee/Sponsor.
4. Severe dyskinesia in the opinion of either the investigator or the Enrollment Approval Committee.
5. Treatment with non-selective monoamine oxidase (MAO) inhibitors during the last 28 days prior to initial screening assessment or planning to take during study participation
6. Previous or planned neurosurgical treatment for Parkinson's Disease (e.g., procedures including ablation or deep brain stimulation) during the course of the study
7. Significant cognitive impairment as defined by the Mini-Mental State Examination (MMSE) score < 26.
8. Clinically significant psychiatric illness, including major depression (Hamilton Depression Rating Scale-17 ≥14). Subjects with a lifetime history of suicidal attempt (including an active attempt, interrupted attempt or aborted attempt)
9. Current or previous treatment for more than 1 month within the past 2 years with any neuroleptic drug (antipsychotic) or any other drug with anti-dopaminergic properties (e.g. metoclopramide, domperidone)
10. Currently experiencing or any known history of psychosis or delusions within 2 years prior to Screening.
11. Known history of substance abuse within the past 2 years
12. Moderate or greater level of alcohol consumption
13. Unable to swallow large pills (e.g., large vitamin pills)
14. History of Melanoma or suspicious skin lesion which could be a Melanoma
15. Narrow-angle Glaucoma
16. History of small bowel or gastric surgery (Including PEG-J placement for Duopa/Duodopa) or bowel obstruction, diagnosis of small bowel narrowing, diagnosis of Crohn's disease, or frequent nausea or emesis, regardless of etiology, (Previous appendectomy or hernioplasty will not be exclusionary).
17. Active peptic ulcer disease or a history of peptic ulcer or upper GI bleeding
18. Regular use of opioids (Intermittent opioid use is not exclusionary)
19. Symptomatic gastroparesis with frequent vomiting (at least once a week)
20. Concomitant use of NSAIDs and oral steroids within the past 28 days
21. Allergy to the study drug or any of its excipients, or to Yellow Dye #5 (tartrazine)
22. Women who are pregnant or nursing. Women of childbearing potential who are not willing to use a medically acceptable method of contraception.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-07 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline through study completion, an average of 27 weeks, in the percentage of daily "Off time" during waking hours | Baseline through study completion, an average of 27 weeks
  Change from Baseline through study completion, an average of 27 weeks, in the percentage of daily "Off time" during waking hours based on Hauser Home Diary assessments; Total number of "Off " hours normalized to a 16- hour waking day will also be calculated but only a single p-value applicable to both the percentage and hours will be reported.

SECONDARY OUTCOMES:
Change from Baseline through study completion, an average of 27 weeks, in "On time" without troublesome dyskinesia during waking hours | Baseline through study completion, an average of 27 weeks
Change in the number of total daily LD doses from Baseline through study completion, an average of 27 weeks (hours) | Baseline through study completion, an average of 27 weeks
CGI-I through study completion, an average of 27 weeks, as recorded by physician & patient | Baseline through through study completion, an average of 27 weeks,
Change from Baseline through study completion, an average of 27 weeks, in total UPDRS Score (Sum of Parts I-III) | Baseline through study completion, an average of 27 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter A LeWitt, MD, Principal Investigator — Henry Ford Hospital - West Bloomfield
Locations (97):
- United States (36):
  - University Alabama Hospital Neurology, Birmingham, Alabama
  - Saint Joseph's Hospital and Medical Center Muhammad Ali Parkinson Research Center, Phoenix, Arizona
  - Parkinson's Disease & Movement Disorders Center, Dept of Neu, Fountain Valley, California
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - SC3 Research, Pasadena, California
  - SC3 Research, Reseda, California
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado Dept. of Neurology, Aurora, Colorado
  - Hartford HealthCare, Vernon, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Collier Neurologic Specialists, LLC, Naples, Florida
  - Bioclinica Research, Orlando, Florida
  - Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - The University of Kansas Hospital, Kansas City, Kansas
  - Boston University School of Medicine, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Henry Ford Hospital, West Bloomfield, Michigan
  - Dartmouth Hitchcock Neurology, Lebanon, New Hampshire
  - Atlantic Health System Hospital Corp.-Overlook Hospital, Summit, New Jersey
  - David L. Kreitzman, MD., PC, Commack, New York
  - Fresco Institute for Parkinson's and Movement Disorders, New York, New York
  - Weill Cornell Medical College of Cornell University, New York, New York
  - Asheville Neurology Specialists, Asheville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Toledo, Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center Vanderbilt Clinical Neurosciences, Nashville, Tennessee
  - North Texas Movement Disorders Institute, Bedford, Texas
  - Baylor College of Medicine Department of Neurology, Houston, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Booth Garner Parkinson's Care Center, Kirkland, Washington
- Bulgaria (5):
  - MHAT 'Sv.Pantaleymon - Pleven' OOD, Pleven
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi" EAD, Plovdiv
  - Clinic for Neurology and Sleep Medicine, Sofia
  - Clinic of Neurological Diseases, Sofia
  - Multiprofile Hospital for Active Treatment "Sveta Marina'' EAD, Varna
- Germany (5):
  - Neuroakademie Alzenau GbR, Aschaffenburg
  - Praxis für Neurologie und Psychiatrie, Berlin
  - Uniklinikum Carl-Gustav Carus an der TU Dresden, Dresden
  - Technischen Universitaet Muenchen (TUM) - Klinikum Rechts der Isar, München
  - Praxis für Neurologie und Psychiatrie, Westerstede
- Israel (4):
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center at Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (12):
  - Ospedale Generale Regionale Francesco Miulli, Acquaviva delle Fonti
  - Ospedali Riuniti di Ancona, Ancona
  - Spedali Civili Di Brescia Azienda Ospedaliera, Brescia
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - IRCCS Neurologico Fondazione "C. Mondino", Pavia
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - IRCCS San Raffaele Pisana, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Universitaria San Giovanni di Dio Ruggi d'Aragona, Salerno
  - Ospedale di Circolo e Fondazione Macchi, Varese
  - Azienda Unitá Locale Socio Sanitaria 12 Veneziana - Ospedale dell'Angelo, Venezia
  - Casa di Cura Villa Margherita, Vicenza
- Poland (8):
  - Centrum Medyczne Damiana Holding, Warsaw, Masovian Voivodeship
  - VITAMED Galaj i Cichomski spólka jawna, Bydgoszcz
  - Anna Kapustecka Prywatna Przychodnia Specjalistyczna STOMED, Częstochowa
  - NEURO-CARE Site Management Organization Gabriela Klodowska-Duda, Katowice
  - Centrum Medyczne Pratia Katowice I, Katowice
  - Krakowska Akademia Neurologii Sp. z o. o., Krakow
  - Gabinet Lekarski Prof. Andrzej Bogucki, Lodz
  - Centrum Medyczne Pratia Warszawa, Warsaw
- Slovakia (3):
  - Neurologicka ambulancia, Euro-Neuro s.r.o., Bratislava
  - KONZÍLIUM s.r.o., Považská Bystrica
  - NEURON - D.T. s.r.o., Žilina
- Spain (10):
  - HM Puerta del Sur, Móstoles, Madrid
  - Hospital Universitari Quirón Dexeus, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Infanta Sofía, San Sebastián de los Reyes
  - Hospital General de Cataluña, Sant Cugat del Vallès
- Ukraine (10):
  - Ukrainian State Scientific Research Institution of Medical and Social Problems of Disability, Cherkasy
  - Dnipropetrovsk medical academy MOH of Ukraine, Dnipro
  - Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine, Kharkiv
  - State Institution "Institute of Gerontology of the AMS of Ukraine", Kyiv
  - Lviv City Clinical Hospital, Lviv
  - Regional Clinical Hospital n.a. N.V. Sklifosovskyi, Poltava
  - Municipal Institution "Zaporizhzhya City Clinical Multidisciplinary Hospital #9", Zaporizhzhya
  - Municipal Institution 6¿ City Clinical Hospital, Zaporizhzhya
  - Clinical Hospital #2, Zaporozh’ye
  - Municipal Institution Zaporizhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporozh’ye
- United Kingdom (4):
  - Fairfield General Hospital, Bury
  - Newcastle University Clinical Ageing Research, Newcastle upon Tyne
  - Queens Medical Centre Nottingham, University Hospital, Nottingham
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS: 1. GENE THERAPY FOR PARKINSON'S, 2. PHASE 3 STUDY IN FOCUS - INTEC PHARMA'S ACCORDION PILL, 3. CLINICAL TRIALS RESOURCES. J Parkinsons Dis. 2019;9(2):251-264. doi: 10.3233/JPD-199001. No abstract available. PMID 31127735